CLINICAL TRIAL: NCT03699618
Title: Anti-VEGF Therapy for Subfoveal Hemorrhage in Patients With Neovascular Age-Related Macular Degeneration
Status: Terminated | Type: Observational
Why Stopped: Challenging Enrollment
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00178395
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Submacular Hemorrhage; Wet Macular Degeneration; Neovascular Age-related Macular Degeneration
Keywords: NVAMD; Anti-VEGF
MeSH Terms: conditions — Wet Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anti-VEGF injection only: Patients who will receive monthly intravitreal anti-VEGF injection for 12 months, followed by anti-VEGF at standard of care treatment interval during months 12-24
  Interventions: Drug: Anti-VEGF
- Hemorrhage displacement + Anti-VEGF: Hemorrhage displacement (at investigators' discretion) followed by monthly intravitreal anti-VEGF injections for 12 months, and standard of care treatment interval during months 12-24
  Interventions: Other: Hemorrhage displacement + Anti-VEGF

INTERVENTIONS:
Drug: Anti-VEGF — Standard of care treatment with anti-VEGF only
  Groups: Anti-VEGF injection only
Other: Hemorrhage displacement + Anti-VEGF — Standard of care treatment with hemorrhage displacement (at investigators' discretion) followed by anti-VEGF injections
  Groups: Hemorrhage displacement + Anti-VEGF

SUMMARY:
This study will define the limits of subretinal hemorrhage parameters that are consistent with a good visual outcome with aggressive anti-VEGF treatment in patients with neovascular age-related macular degeneration (NVAMD).

DETAILED DESCRIPTION:
The purpose of this study is to define the limits of subretinal hemorrhage parameters that are consistent with a good visual outcome with aggressive anti-vascular endothelial growth factor (anti-VEGF) treatment, thereby providing guidance as to when it is reasonable to treat with anti-VEGF and when it is necessary to displace the hemorrhage in addition to treating with anti-VEGF.

This is a prospective study that will enroll 98 patients with subretinal hemorrhage in the fovea [also known as subfoveal hemorrhage (SFH)] secondary to neovascular AMD at the Wilmer Eye Institute, Johns Hopkins Hospital (Downtown campus and all other Eye Care Network clinics). The primary endpoint is at month 12 and the secondary endpoint is at month 24. The duration of the study is 24 months.

Study visits will include a baseline visit, then monthly visits for 12 months, followed by standard care treatment visits in the second year until month 24. The patients will be stratified into two groups based on standard of care management: 1. Patients receiving intravitreal (IVT) anti-VEGF injections; 2. Patients undergoing SFH displacement followed by IVT anti-VEGF injections. Patients will receive monthly anti-VEGF injection for 12 months, followed by anti-VEGF at standard of care treatment interval during months 12-24; or SFH displacement (at investigators' discretion) followed by monthly IVT anti-VEGF injections for 12 months, and standard of care treatment interval during months 12-24.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and authorization of use and disclosure of protected health information
* Age 50 years or older
* Presence of subretinal hemorrhage (SRH) involving the fovea in patients with NVAMD including polypoidal choroidal vasculopathy (PCV)

Exclusion Criteria:

* SFH in the study eye due to causes other than NVAMD
* Media opacity due to concurrent vitreous hemorrhage or cataracts that preclude adequate imaging
* Substantial loss of VA due to condition other than AMD
* Limited visual potential from substantial atrophy or fibrosis in fovea
* Poor visual potential with known permanent reduction in visual acuity prior to SFH

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who develop subretinal hemorrhage (SRH) involving the fovea secondary to neovascular age-related macular degeneration will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Correlation between hemorrhage characteristics and good visual outcome at month 12 | 12 months
  Correlation between baseline SFH characteristics measured on Spectralis SD-OCT (size and thickness of SFH, and shortest distance between border of SFH and fovea) and good visual acuity outcome (≥20/50) after controlling for baseline visual acuity in patients receiving monthly IVT anti-VEGF injections using pearson or spearman correlation coefficients based on normality of the data.

SECONDARY OUTCOMES:
Correlation between hemorrhage characteristics and visual acuity at month 12 | 12 months
  Correlation between baseline SFH characteristics measured on Spectralis SD-OCT (size and thickness of SFH, and shortest distance between border of SFH and fovea) and VA at 12-months using linear regression model accounting for all clinically relevant covariates including baseline VA
Correlation between hemorrhage characteristics and visual acuity at month 24 | 24 months
  Correlation between baseline SFH characteristics measured on Spectralis SD-OCT (size and thickness of SFH, and shortest distance between border of SFH and fovea) and VA at 24-months using linear regression model accounting for all clinically relevant covariates including baseline VA
Correlation between hemorrhage characteristics and good visual outcome at month 24 | 24 months
  Correlation between baseline SFH characteristics measured on Spectralis SD-OCT (size and thickness of SFH, and shortest distance between border of SFH and fovea) and good visual acuity outcome (≥20/50) after controlling for baseline visual acuity in patients receiving monthly IVT anti-VEGF injections using pearson or spearman correlation coefficients based on normality of the data.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Campochiaro, MD, Principal Investigator — Wilmer Eye Institute
Locations (1):
- Wilmer Eye Institute, Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kherani S, Scott AW, Wenick AS, Zimmer-Galler I, Brady CJ, Sodhi A, Meyerle C, Solomon SD, Shaukat R, Channa R, Adeyemo O, Handa JT, Wang J, Campochiaro PA. Shortest Distance From Fovea to Subfoveal Hemorrhage Border Is Important in Patients With Neovascular Age-related Macular Degeneration. Am J Ophthalmol. 2018 May;189:86-95. doi: 10.1016/j.ajo.2018.02.015. Epub 2018 Feb 28. PMID 29499174
- [Background] Iacono P, Parodi MB, Introini U, La Spina C, Varano M, Bandello F. Intravitreal ranibizumab for choroidal neovascularization with large submacular hemorrhage in age-related macular degeneration. Retina. 2014 Feb;34(2):281-7. doi: 10.1097/IAE.0b013e3182979e33. PMID 23851632
- [Background] Kim JH, Chang YS, Kim JW, Kim CG, Yoo SJ, Cho HJ. Intravitreal anti-vascular endothelial growth factor for submacular hemorrhage from choroidal neovascularization. Ophthalmology. 2014 Apr;121(4):926-35. doi: 10.1016/j.ophtha.2013.11.004. Epub 2013 Dec 15. PMID 24342019
- [Background] Kim HS, Cho HJ, Yoo SG, Kim JH, Han JI, Lee TG, Kim JW. Intravitreal anti-vascular endothelial growth factor monotherapy for large submacular hemorrhage secondary to neovascular age-related macular degeneration. Eye (Lond). 2015 Sep;29(9):1141-51. doi: 10.1038/eye.2015.131. Epub 2015 Aug 14. PMID 26272443
- [Background] Shienbaum G, Garcia Filho CA, Flynn HW Jr, Nunes RP, Smiddy WE, Rosenfeld PJ. Management of submacular hemorrhage secondary to neovascular age-related macular degeneration with anti-vascular endothelial growth factor monotherapy. Am J Ophthalmol. 2013 Jun;155(6):1009-13. doi: 10.1016/j.ajo.2013.01.012. Epub 2013 Mar 7. PMID 23465269
- [Background] Altaweel MM, Daniel E, Martin DF, Mittra RA, Grunwald JE, Lai MM, Melamud A, Morse LS, Huang J, Ferris FL 3rd, Fine SL, Maguire MG; Comparison of Age-related Macular Degeneration Treatments Trials (CATT) Research Group; Comparison of Age-related Macular Degeneration Treatments Trials CATT Research Group. Outcomes of eyes with lesions composed of >50% blood in the Comparison of Age-related Macular Degeneration Treatments Trials (CATT). Ophthalmology. 2015 Feb;122(2):391-398.e5. doi: 10.1016/j.ophtha.2014.08.020. Epub 2014 Oct 11. PMID 25307130
- [Background] Treumer F, Roider J, Hillenkamp J. Long-term outcome of subretinal coapplication of rtPA and bevacizumab followed by repeated intravitreal anti-VEGF injections for neovascular AMD with submacular haemorrhage. Br J Ophthalmol. 2012 May;96(5):708-13. doi: 10.1136/bjophthalmol-2011-300655. Epub 2011 Dec 15. PMID 22174095